CLINICAL TRIAL: NCT04508868
Title: Behavioral Activation and Mental Imagery Delivered Via Telephone for the Treatment of Depressive Symptoms in Older Individuals in Isolation During Covid-19: A Randomized Clinical Trial
Brief Title: Treatment of Depressive Symptoms in Older Individuals in Isolation During Covid-19
Acronym: CoviDep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to changes in government restrictions. Collected data to be presented as a pilot study.
Sponsor: Uppsala University (Other)
Collaborators: Västmanland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02079
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Depression; Depressive Symptoms
Keywords: Depression; Depressive Symptoms; Cognitive Behavioral Therapy; Social Isolation; Coronavirus; Pandemic
MeSH Terms: conditions — Depression; Social Isolation; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Activation with Mental Imagery (Experimental): Four weekly sessions of Brief Behavioral Activation with Mental Imagery.
  Interventions: Behavioral: Brief Behavioral Activation with Mental Imagery
- Minimal Attention Control Intervention (Placebo Comparator): Four weeks with weekly follow-up calls.
  Interventions: Behavioral: Minimal Attention Control Intervention

INTERVENTIONS:
Behavioral: Brief Behavioral Activation with Mental Imagery — Session 1:
  Provide psychoeducation about depression; Provide treatment rationale for BA; Provide rationale and instructions for activity log; Plan activities for coming week.
  Session 2:
  Review activity log; Discuss life goals and values; Plan activities aligned with life goals and values for coming week; Provide rationale for Mental Imagery (MI); Go through MI-exercise for one of the planned activities.
  Session 3:
  Review activity log; Troubleshoot any problems carrying out activities; Plan activities aligned with life goals and values for coming week; Go through MI-exercise for one of the planned activities.
  Session 4:
  Review activity log; Troubleshoot any problems carrying out activities; Review treatment; Stress the importance of continuing to engage in activities aligned with life goals and values; Referral to additional services if necessary.
  Arms: Brief Behavioral Activation with Mental Imagery
Behavioral: Minimal Attention Control Intervention — Weekly call with follow-up of psychiatric symptoms and assessment of suicide risk.
  Arms: Minimal Attention Control Intervention

SUMMARY:
This research study is designed to investigate the effects of a brief psychological intervention for improving depressed mood in older individuals (65 years and older) in isolation during the Coronavirus (COVID-19) pandemic. The treatment is delivered by telephone and consists of four weekly individual sessions. Two therapeutic methods are used in combination during this intervention: Behavioral activation (BA) and Mental Imagery (MI). BA involves identifying and scheduling enjoyable and meaningful activities to improve mood and reduce social isolation. To enhance BA efficacy and adherence, MI is paired with BA as MI is known to activate emotion and motivation. The MI intervention in this study involves having participants imagine, in vivid sensory detail, engaging in some of the activities that are scheduled during BA.

Approximately 154 individuals will participate in the study. Half of the participants will be randomised to start the intervention immediately, while the other half of the participants will be randomized to a control group receiving the intervention after 4 weeks. This procedure makes it possible to evaluate the effects of the treatment while not disadvantaging participants randomized to the control group. Participants will be asked to fill in questionnaires before, during (at the end of each intervention week), and after treatment (or waiting period for the control group). Questionnaires will also be sent 1-, 3- and 6 months after treatment to follow up on the results. A smaller group of participants (10-15) will be asked to participate in a more detailed interview about how they experienced the treatment.

DETAILED DESCRIPTION:
Coronavirus (COVID-19) has become a worldwide pandemic. The mortality rates are highest in the older age groups, particularly in those 70 years and older. In Sweden, the government urges people 70 years and older to limit close contact with other people and to stay at home as much as possible, a strategy called social distancing. From previous epidemics, such as the SARS-epidemic, we know that quarantine and isolation leads to psychological symptoms such as stress, irritability, depressed mood and sleep problems. About 30% of those subjected to isolation and quarantine become depressed, and in a study from Hong Kong during SARS there was a nearly 32% increase of suicide rates among individuals 65 years and older. In Sweden, depression among the elderly was a major public health concern before the covid-19-pandemic - Major depression occurred in 5-15 % of the older population in Sweden, and one third of the women and a fifth of the men 65 years and older reported subclinical depressive symptoms. Several mental health experts raise concerns that there will be an increase of psychiatric illness during and after covid-19, particularly among the elderly.

Depression in older individuals can be treated with antidepressant medication, psychological interventions and physical activity. However, the majority of the older individuals state that they would prefer psychological treatments to medication, which poses a challenge during COVID-19 as such treatments are often delivered face-to-face. Psychological treatments delivered via the Internet are as efficacious as face-to-face, but only 3-4% of the individuals 65 years and above in Sweden use digital applications that replace physical healthcare visits.

Psychological treatments have been shown to work when delivered via telephone, and since practically every household in Sweden has access to a telephone, the investigators believe this could be a feasible option. Preferably, the treatment should be brief yet effective, and easily accessible for healthcare professionals. One such treatment is brief behavioral activation (BA), which is aimed at increasing enjoyable and meaningful activities to improve mood. BA has been shown to be feasible in as few as four sessions. Depression is often accompanied by low motivation and lack of energy, which can pose a problem when trying to increase activities. One way of increasing motivation in BA and the likelihood of performing the planned activities is to add mental imagery (MI), where some of these activities are imagined in detail during the calls.

However, there are to the investigators knowledge no studies of telephone-delivered brief BA for older individuals, no studies of the combination of BA and MI for depression in the elderly, and no studies of either of these during pandemics with isolation or quarantine.

The aim of the present study is to investigate the feasibility, effect and experience of telephone-delivered Behavioral Activation with Mental Imagery for the treatment of depressive symptoms in individuals 65 years and older during the covid-19-pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the County of Västmanland
* Access to telephone
* Fluent in written and spoken Swedish
* Reporting clinically significant depressive symptoms above cut-of on depression measures and/or by structured clinical interview

Exclusion Criteria:

* Severe depression
* Elevated risk of suicide
* Current substance use disorder
* Current or previous manic/hypomanic episodes
* Current psychotic disorder
* Current diagnosis of dementia/major neurocognitive disorder
* Currently receiving psychological therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms using the Montgomery-Asberg Depression Rating Scale, MADRS-S | Baseline; Intervention Week 1; Intervention Week 2; Intervention Week 3; Intervention Week 4; 1 month post-intervention; 3 months post-intervention; 6 months post-intervention.
  MADRS-S is a nine-item questionnaire used to measure severity of depression. The score ranges from 0-54.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms using the Geriatric Depression Rating Scale 15, GDS-15 | Baseline; Intervention Week 4; 1 month post-intervention; 3 months post-intervention; 6 months post-intervention.
  GDS-15 is a 15-item questionnaire used to identify depression in the elderly. The score ranges from 0-15.
Change from baseline in depressive symptoms using the Patient Health Questionnaire 9, PHQ-9 | Baseline; Intervention Week 4; 1 month post-intervention; 3 months post-intervention; 6 months post-intervention.
  PHQ-9 is a nine-item questionnaire used to identify depression as well as measuring severity of depression. The score ranges from 0-27.
Change in depression diagnosis assessed using the Mini International Neuropsychiatric Interview, MINI | Baseline; Intervention Week 4.
  MINI is a structured clinical interview used to assess the presence/absence of common psychiatric disorders.
Change from baseline in anxiety symptoms using the Generalized Anxiety Disorder 7-item, GAD-7 | Baseline; Intervention Week 4; 1 month post-intervention; 3 months post-intervention; 6 months post-intervention.
  GAD-7 is a seven-item questionnaire used to identify generalized anxiety disorder as well as measuring severity of anxiety symptoms. The score ranges from 0-21.
Change from baseline in behavioral activation using The Behavioral Activation for Depression Scale - Short Form, BADS-SF | Baseline; Intervention Week 4; 1 month post-intervention; 3 months post-intervention; 6 months post-intervention.
  BADS-SF is a nine-item questionnaire used to measure changes in avoidance and activation. The score ranges from 0-54.
Change from baseline in health and disability using The WHO Disability Assessment Schedule 12-item, WHODAS | Baseline; Intervention Week 4; 1 month post-intervention; 3 months post-intervention; 6 months post-intervention.
  WHODAS-12 is a 12-item questionnaire used to assess disability due to health conditions. The total score ranges from 0-48.
Adverse and unwanted effects of the experimental intervention using the Negative Effects Questionnaire, NEQ | Experimental Intervention Week 4.
  NEQ is a 20-item questionnaire used to assess adverse and unwanted effects of psychological treatments.
Mental imagery is assessed at baseline using the Plymouth Sensory Imagery Questionnaire, Psi-Q | Baseline; Intervention Week 4.
  Psi-Q is a 35-item questionnaire assessing the vividness of mental imagery. In this study we plan to use the visual subscale with five items, with a total score ranging from 0-50.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Damberg, MD, PhD, Principal Investigator — County of Vastmanland and Uppsala University
Locations (1):
- Adult Psychiatric Clinic, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified outcome measure IPD will be shared upon reasonable requests from academic researchers.
Supporting Information: Study Protocol, SAP
Time Frame: * Study protocol to be shared before data collection is completed
  * Statistical Analysis Plan to be shared before data analysis begin
Access Criteria: Data will be shared upon reasonable requests assessed by the investigators.